CLINICAL TRIAL: NCT05867836
Title: Trial of Adherence and Acceptance of Multiple Micronutrient Supplementation (MMS) vs Iron and Folic Acid (IFA) Among Pregnant Women and Health System Enablers and Constraints Related to MMS in Cambodia
Brief Title: Multiple Micronutrient Supplementation vs Iron and Folic Acid Among Pregnant Women in Cambodia
Acronym: MMS-Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Helen Keller International (Other); Vitamin Angels (Unknown)
Responsible Party: Principal Investigator, Crystal Karakochuk, Assistant Professor, Human Nutrition, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H23-01316
Record Dates: First submitted 2023-04-24; First posted 2023-05-22 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Related; Antenatal Care; Iron Folic Acid Supplementation
Keywords: Multiple micronutrient supplementation; Adherence; Acceptability

STUDY DESIGN:
Intervention Model Description: Clinical trial to assess the adherence and acceptability of iron and folic acid (IFA) vs. multiple micronutrient supplementation (MMS) during pregnancy in Cambodian women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IFA-90 (Active Comparator): Iron and folic acid (IFA) for 90 days
  Interventions: Dietary Supplement: IFA vs. MMS during pregnancy
- MMS-90 (Experimental): Multiple micronutrient supplementation (MMS) for 90 days with 2 distributions of MMS supplements (2 x 90 pill bottles; distributed at different ANC visits)
  Interventions: Dietary Supplement: IFA vs. MMS during pregnancy
- MMS-180 (Experimental): Multiple micronutrient supplementation (MMS) for 180 days but with 1 distribution of MMS supplements (1 x 180 pill bottle)
  Interventions: Dietary Supplement: IFA vs. MMS during pregnancy

INTERVENTIONS:
Dietary Supplement: IFA vs. MMS during pregnancy — Iron and folic acid, or multiple micronutrient supplements provided during pregnancy

SUMMARY:
Iron and folic acid (IFA) supplements are currently provided to Cambodian women during pregnancy. However, recent research has showed benefit of a multiple micronutrient supplement (MMS) over just IFA alone on several outcomes of perinatal and infant health. The Ministry of Health in Cambodia has proposed a transition from IFA to MMS but would like to collect some formative research on this first to assess acceptability and adherence to MMS (over IFA) and help guide key messaging, packaging, and practices to guide the transition in Cambodia.

DETAILED DESCRIPTION:
Antenatal multiple micronutrient supplementation (MMS) is a potentially cost-effective, scalable approach that can contribute to addressing the persistent challenge of maternal undernutrition, reducing low birth weight, reducing small-for-gestational age births, and potentially reducing preterm birth. A 2019 independent patient (IDP) meta-analysis indicates MMS decreased mortality for female neonates and provided greater reductions in the risk of low birthweight and preterm birth for infants born to undernourished and anemic women. The 2019 Cochrane Review compared the effects of MMS to iron folic acid (IFA) supplementation in another review and meta-analysis and found MMS supplementation was associated with reduced small-for-gestational age births. Operationalizing MMS interventions in different country contexts is urgently needed to improve the health of mothers and children. However, guidelines on antenatal MMS supplementation have yet to be widely adopted into national policies, in part because the WHO guidelines do not reflect recent evidence.

Helen Keller Intl, with support from Vitamin Angels, conducted a landscape analysis of antenatal MMS supplementation in Cambodia to supportive or potentially supportive stakeholders to accelerate MMS uptake and use in Cambodia. During a stakeholder consultation help in September 2021, workshop participants concluded it is an appropriate time to consider the transition from iron folic acid supplementation (IFA) to MMS supplementation. Following this consultation, a multi-stakeholder Steering Committee was formed, consisting of technical and government representatives from a range of disciplines, to oversee and support this transition.

The landscape analysis revealed that key Cambodian stakeholders are open to exploring the feasibility of a transition from IFA to MMS supplementation for pregnant women and identified key operational and implementation research priorities to inform the transition process. One of those questions relates to the acceptability by pregnant women of MMS in terms of packaging, color, ease of consumption, taste, and overall liking.

The landscape analysis also highlighted the need to assess the adherence of MMS vs. IFA supplementation. WHO recommends that all pregnant women receive a standard dose of 30-60 mg iron and 400 µg folic acid beginning as soon as possible during pregnancy. Ideally, women should receive IFA no later than the first trimester of pregnancy, which means taking 180 tablets before delivery. It is important to note that many countries (including Cambodia) aim for women to receive 90 or more tablets during pregnancy. Currently, in Cambodia the government is distributing 90 tablets of IFA to pregnant women attending public antenatal care services. Thus, to transition from 90 tablets of IFA to 180 tablets is not as easy as a pill switch. To ensure pregnant women can receive the full benefits from MMS supplementation, transitioning from IFA to MMS will require pregnant women to come into ANC during their first trimester and adhere to the recommended 180 tablets of MMS throughout their pregnancy.

To date there are no published studies or documentation from Cambodia on pregnant women's acceptability of MMS supplements or adherence to a 180-dosage regimen of MMS. A 2011 study in two provinces in Cambodia found access to antenatal care (ANC), the number of supplements provided, and ANC attendance were the strongest determinants for adherence to IFA supplementation. Another analysis in Cambodia found the primary reasons for not taking the WHO recommended number of 180 IFA doses (WHO, 2012) were starting ANC after the 1st trimester and not attending all recommended ANC visits. In Nepal, researchers have found knowledge about preventable conditions and benefits, perceived barriers, social support, and perceived severity of not taking the supplement predicted IFA compliance while other also found forgetting to take the supplements was a barrier. In a study from Vietnam, determinants of adherence to either folic acid, IFA, or MMS supplementation were socioeconomic status, ethnicity, occupation, and parity, as well as increased contact with health workers. Acceptability studies which included MMS supplementation have identified organoleptic properties perceived benefits, and fears or perceived negative effects as influential factors on acceptance and utilization.

Following the landscape analysis, Vitamin Angels and Helen Keller co-hosted with the Ministry of Health (MoH) a Consensus Building Stakeholder Workshop. Workshop participants recommended conducting a pilot test to engage with the pregnant women who are going to be consuming the product, as well as with the health care actors who will be involved in product delivery. Following the workshop, the MoH formed an MMS Steering Committee comprised of many key stakeholders within the MoH, United Nations, and civil society. The MMS Steering Committee will review the implementation research protocol, provide guidance, and, also, meet quarterly to review implementation progress and feedback on development of health provider counseling materials and other strategic behavioral change materials.

Assessment of the acceptability and feasibility of a new intervention should be done with end users prior to implementation, especially when the strategy requires possible changes in care processes. Determining the acceptability of MMS supplements with pregnant women will enhance understanding of barriers to implementation and help to develop an MMS supplementation scale-up strategy that is feasible and cost-effective. Implementation strategies will need to consider a host of drivers that influence acceptability and adherence, including MMS product availability, affordability, and acceptability as well as improvements to health seeking behaviors during pregnancy. Determining non-inferiority of adherence is also critical when introducing a new supplement. Given the dearth of studies and knowledge around MMS supplementation in Cambodia, Helen Keller and Vitamin Angels propose formative and implementation research to identify factors influencing adherence to antenatal supplementation to effectively inform an MMS supplementation strategy and ANC service delivery.

Rationale for the Study MMS supplements are a new product for pregnant women and health providers in Cambodia. As it is intended to replace IFA, MMS supplementation uptake requires careful introduction and transition to ensure optimal supplement acceptability and compliance, without which improving maternal nutrition may remain a challenge. As others have suggested that transitioning to MMS therefore requires a formative research phase to inform programming and service delivery. Specifically, testing product acceptability, labeling, packaging, health worker capacity building strategies, and behavioral change messaging to promote daily use among Cambodian pregnant women is important before fully transitioning to and scaling up MMS supplementation. Furthermore, concerns expressed by host-country stakeholders question the impact on ANC use (ensuring at least four visits) if MMS is provided in a large quantity (i.e., 90 or 180 tablets) to pregnant women need to be explored.

Aim and Objectives The aim of this study is to assess factors that influence optimal MMS consumption, defined as 180 tablets during pregnancy, and provide recommendations to the MoH MMS Steering Committee to effectively transition to distribution of 180 tablets of MMS supplements as part of routine ANC services. Specific recommendations generated by this study will be related to product acceptability, packaging, labeling, training needs, behavioral change messaging, adherence, and best ways to integrate MMS within ANC services. Results of this adherence research are intended to be used by the MoH and the MMS Steering Committee.

This study has the following objectives:

1. Assess acceptability of IFA and MMS supplements.
2. Assess adherence to recommended IFA and MMS supplementation.
3. Assess non-inferiority of MMS compared to IFA supplementation.
4. Assess impact of pill quantity provided at one time on ANC attendance.
5. Evaluate factors that influence adherence behavior.
6. Develop recommendations for product marketing and service delivery to encourage adherence to MMS supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Age 18-45 years
* Gestational age less than 14 weeks
* Low risk pregnancy
* Live in Kampong Thom and will not move away within the next 6 months
* Agree to have data collectors come to your home once a month to complete a survey and pill weighing or counting

Exclusion Criteria:

* Women participating in any nutrition programs beyond the normal care provided though government facilities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1545 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Adherence (counts) | 90 days for the IFA-90 group and 180 days for the MMS-180 group
  Adherence as per pill count at the final visit

SECONDARY OUTCOMES:
Adherence (weights) | 90 days for the IFA-90 group and 180 days for the MMS-180 group
  Adherence as per pill weight (g) at the final visit
Acceptability (quantitative) | 30 day-, 90 day- and 180-day timepoints
  Acceptability as per survey questionnaire
Acceptability (qualitative) | 90 days for IFA group and 180 days for MMS-180 group
  Acceptability as per informant interviews

CONTACTS AND LOCATIONS:
Overall Officials: Hou Kroeun, Study Director — Helen Keller International; Crystal D Karakochuk, Principal Investigator — University of British Columbia; Mai A Hoang, Study Director — Helen Keller International
Locations (1):
- Kampong Thom province, Kampong Thom, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clermont A, Kodish SR, Matar Seck A, Salifou A, Rosen J, Grais RF, Isanaka S. Acceptability and Utilization of Three Nutritional Supplements during Pregnancy: Findings from a Longitudinal, Mixed-Methods Study in Niger. Nutrients. 2018 Aug 12;10(8):1073. doi: 10.3390/nu10081073. PMID 30103529
- [Background] Gonzalez-Casanova I, Nguyen PH, Young MF, Harding KB, Reinhart G, Nguyen H, Nechitillo M, Truong TV, Pham H, Nguyen S, Neufeld LM, Martorell R, Ramakrishnan U. Predictors of adherence to micronutrient supplementation before and during pregnancy in Vietnam. BMC Public Health. 2017 May 16;17(1):452. doi: 10.1186/s12889-017-4379-4. PMID 28511688
- [Background] Gupta P, Ray M, Dua T, Radhakrishnan G, Kumar R, Sachdev HP. Multimicronutrient supplementation for undernourished pregnant women and the birth size of their offspring: a double-blind, randomized, placebo-controlled trial. Arch Pediatr Adolesc Med. 2007 Jan;161(1):58-64. doi: 10.1001/archpedi.161.1.58. PMID 17199068
- [Background] Keats EC, Haider BA, Tam E, Bhutta ZA. Multiple-micronutrient supplementation for women during pregnancy. Cochrane Database Syst Rev. 2019 Mar 14;3(3):CD004905. doi: 10.1002/14651858.CD004905.pub6. PMID 30873598
- [Background] Kulkarni B, Christian P, LeClerq SC, Khatry SK. Determinants of compliance to antenatal micronutrient supplementation and women's perceptions of supplement use in rural Nepal. Public Health Nutr. 2010 Jan;13(1):82-90. doi: 10.1017/S1368980009005862. Epub 2009 May 19. PMID 19454124
- [Background] Lacerte P, Pradipasen M, Temcharoen P, Imamee N, Vorapongsathorn T. Determinants of adherence to iron/folate supplementation during pregnancy in two provinces in Cambodia. Asia Pac J Public Health. 2011 May;23(3):315-23. doi: 10.1177/1010539511403133. PMID 21593006
- [Background] Smith ER, Shankar AH, Wu LS, Aboud S, Adu-Afarwuah S, Ali H, Agustina R, Arifeen S, Ashorn P, Bhutta ZA, Christian P, Devakumar D, Dewey KG, Friis H, Gomo E, Gupta P, Kaestel P, Kolsteren P, Lanou H, Maleta K, Mamadoultaibou A, Msamanga G, Osrin D, Persson LA, Ramakrishnan U, Rivera JA, Rizvi A, Sachdev HPS, Urassa W, West KP Jr, Zagre N, Zeng L, Zhu Z, Fawzi WW, Sudfeld CR. Modifiers of the effect of maternal multiple micronutrient supplementation on stillbirth, birth outcomes, and infant mortality: a meta-analysis of individual patient data from 17 randomised trials in low-income and middle-income countries. Lancet Glob Health. 2017 Nov;5(11):e1090-e1100. doi: 10.1016/S2214-109X(17)30371-6. PMID 29025632
- [Background] Sudfeld CR, Smith ER. New Evidence Should Inform WHO Guidelines on Multiple Micronutrient Supplementation in Pregnancy. J Nutr. 2019 Mar 1;149(3):359-361. doi: 10.1093/jn/nxy279. PMID 30773589
- [Background] Young SL, Blanco I, Hernandez-Cordero S, Pelto GH, Neufeld LM. Organoleptic properties, ease of use, and perceived health effects are determinants of acceptability of micronutrient supplements among poor Mexican women. J Nutr. 2010 Mar;140(3):605-11. doi: 10.3945/jn.109.113498. Epub 2010 Jan 27. PMID 20107141
- [Background] West KP Jr, Shamim AA, Mehra S, Labrique AB, Ali H, Shaikh S, Klemm RD, Wu LS, Mitra M, Haque R, Hanif AA, Massie AB, Merrill RD, Schulze KJ, Christian P. Effect of maternal multiple micronutrient vs iron-folic acid supplementation on infant mortality and adverse birth outcomes in rural Bangladesh: the JiVitA-3 randomized trial. JAMA. 2014 Dec 24-31;312(24):2649-58. doi: 10.1001/jama.2014.16819. PMID 25536256
- [Derived] Sauer C, Hoang MA, Kroeun H, Gupta AS, Ngik R, Sokchea M, Labonte JM, Chea M, Klemm R, Mishra A, Panicker A, Sokhal V, Karakochuk CD. Assessing the adherence and acceptability to iron and folic acid compared with multiple micronutrient supplements during pregnancy: a cluster-randomized noninferiority trial in Cambodia. Am J Clin Nutr. 2025 Jul;122(1):166-173. doi: 10.1016/j.ajcnut.2025.04.033. Epub 2025 May 5. PMID 40334750
- [Derived] Hoang MA, Kroeun H, Klemm R, Gupta AS, Rem N, Meng S, Prak S, Rattana K, Chea M, Karakochuk CD, Sauer C, Mishra A, Mohan D, de-Graffenried MJ. Adherence and acceptability of multiple micronutrient supplementation during pregnancy: Study protocol for a cluster-randomized non-inferiority trial in Cambodia. Trials. 2024 Apr 29;25(1):289. doi: 10.1186/s13063-023-07891-z. PMID 38685109